CLINICAL TRIAL: NCT03300557
Title: Pilot Study of Daily Exemestane in Women With Complex Atypical Hyperplasia of the Endometrium/Endometrial Intraepithelial Neoplasia or Low Grade Endometrial Cancer
Brief Title: Exemestane in Treating Patients With Complex Atypical Hyperplasia of the Endometrium/Endometrial Intraepithelial Neoplasia or Low Grade Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2017-01782; NCI-2017-01782 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UW17010; N01-CN-2012-00033; 2016LS183 / UWI17010/UAB1788 (Other: University of Wisconsin Carbone Cancer Center - University Hospital); UWI2016-08-01 (Other: DCP); N01CN00033 (NIH); P30CA014520 (NIH)
Record Dates: First submitted 2017-10-02; First posted 2017-10-03 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Atypical Hyperplasia; Endometrial Atypical Hyperplasia/Endometrioid Intraepithelial Neoplasia; Endometrial Carcinoma; FIGO Grade 1 Endometrial Endometrioid Adenocarcinoma; FIGO Grade 2 Endometrial Endometrioid Adenocarcinoma
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms | interventions — exemestane; Pharmacogenomic Variants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (exemestane) (Experimental): Patients receive exemestane PO QD over 21-42 days in the absence of disease progression or unaccepted toxicity. Patients undergo standard of care surgery between days 22-43.
  Interventions: Drug: Exemestane; Other: Laboratory Biomarker Analysis; Other: Pharmacokinetic Study; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Exemestane — Given PO
  Other Names: Aromasin; FCE-24304
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacokinetic Study — Correlative studies
  Other Names: PHARMACOKINETIC; PK Study
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot phase IIa trial studies how well exemestane works in treating patients with complex atypical hyperplasia of the endometrium/endometrial intraepithelial neoplasia or low grade endometrial cancer. Exemestane may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if there is a decrease in proliferation index, measured by Ki-67 expression, in complex atypical hyperplasia (CAH)/endometrial intraepithelial neoplasia (EIN) or low grade (grade 1 and grade 2) endometrial cancer cells from baseline to post-exemestane treatment.

SECONDARY OBJECTIVES:

I. Circulating serum estradiol and progesterone. II. Pathological response (regression of CAH/EIN or low grade [grade 1 and grade 2] endometrial carcinoma).

III. Tissue biomarkers. IV. Deoxyribonucleic acid (DNA) mutational analysis through next generation sequencing and methylation status of endometrial tumor.

V. Protein markers via tampon recovery before and after treatment. VI. DNA markers via tampon recovery. VII. Safety and adverse effects of treatment. VIII. Comparison of Ki-67 expression changes between study subjects and a historical cohort.

IX. Evaluation of the levels of exemestane in the plasma samples pre and post treatment.

OUTLINE:

Patients receive exemestane orally (PO) once daily (QD) over 21-42 days in the absence of disease progression or unaccepted toxicity. Patients undergo standard of care surgery between days 22-43.

After completion of study treatment, patients with unresolved adverse events on day of surgery are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Females with a histologically proven CAH/ EIN or low grade (grade 1 or grade 2) endometrial carcinoma (EC) for which surgery is planned; the pathologic report from the referring facility will be used to determine pathologic eligibility; this report must be within 45 days of their baseline (pre-surgical) clinic visit
* No prior treatment for CAH/EIN/EC
* Post-menopausal confirmed with one the following criteria:

  * >= 60 years of age
  * Age 56 to 59 years of age with >= 2 years of amenorrhea
  * Age 56 to 59 years of age with < 2 years of amenorrhea and follicle stimulating hormone (FSH) within institutional post-menopausal range.
  * Age 45 to 55 years of age with FSH within institutional post-menopausal range. The Ki-67 expression changes based on menopausal status and specifically varies based on what phase of the menstrual cycle the sample is collected. Therefore, in order to eliminate this source of variability, only postmenopausal women will be included in this trial. In addition, exemestane is currently approved for use in post-menopausal women only.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Hemoglobin >= 9 g/dL
* Serum creatinine =< 1.5 x upper limit of normal or calculated creatinine clearance >= 60 mL/min using Cockcroft-Gault equation for patients with creatinine levels > 1.5 x institutional upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< 1 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* White blood cell (WBC) >= 3000/mcl
* Platelets >= 100,000/mcl
* Able and willing to take oral medications
* Ability to understand and the willingness to sign a written informed consent document
* Body mass index (BMI) > 20

Exclusion Criteria:

* Participants who had curatively treated invasive malignancies for which all treatments ended within 1 year prior to the study (with the exception of basal cell or squamous cell carcinoma of the skin)
* Not a surgical candidate or surgery is not scheduled within 43 days from starting the study drug
* Receiving any other investigational agents
* Any gastrointestinal condition causing malabsorption or obstruction (e.g. celiac sprue, gastric bypass surgery, strictures, adhesions, history of small bowel resection, blind loop syndrome)
* Has been on any hormonal treatment (including progestin-containing intrauterine device [IUD]) for CAH/EIN or low grade (grade 1 or grade 2) endometrial carcinoma in last 3 months
* Use hormone replacement therapy (including systemic or topical estrogen, progesterone, or testosterone based medication) or/and phytoestrogen supplements (i.e. black cohosh) or has been on progestin (including progestin containing IUD), tamoxifen or aromatase inhibitor within the prior 3 months
* Concomitant use of strong CYP3A4 inducers such as rifampicin, phenytoin, carbamazepine, phenobarbital or St. John's wort as these may significantly reduce the availability of exemestane
* Known hypersensitivity to exemestane or its excipients
* Known intercurrent illness or psychiatric illness/social situations that will limit compliance with study requirements
* Evidence or high suspicion of metastatic disease at enrollment
* Women with severe bone density issues/osteoporosis (defined as any medical treatment for osteoporosis, and/or a T-score of -2.5 or lower, and/or history of fracture of the hip or spine)
* Unwilling or unable to undergo research biopsy during the baseline (pre-surgical) clinic visit, or inadequate research biopsy obtained during the baseline (pre-surgical) clinic visit (determined by the gynecologic oncologist at the time of the subject's pelvic exam)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2025-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Britt K Erickson, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We are aware that CTRP lists 46 as enrollment. PRS shall remain as 40 because: "Potential participants who are screened for the purpose of determining eligibility for the study, but do not participate in the study, are not considered enrolled." Thus, 40 is the proper number because the other 6 were screened and found ineligible, therefore not considered enrolled.
Period: Overall Study
Arm/Group | Treatment (Exemestane)
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Exemestane)
Number analyzed (Participants) | 40
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 13
  60-69 years | 18
  70-79 years | 7
  Unknown | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumor Proliferation
Description: Will be measured by change in Ki-67 expression. Will evaluate the change from baseline to post-exposure in absolute change in percent Ki-67 using one-sample Student's t-test or Wilcoxon signed-rank test, as appropriate.
Time Frame: Baseline up to 2 months
Population: There was not enough tissue to analyze from the other two participants
Measure: Mean (Standard Deviation); unit: percent (represented by mean) of cells
Arm/Group | Treatment (Exemestane)
Number analyzed (Participants) | 38
percent (represented by mean) of cells | -0.17 (0.22)

2. Secondary Outcome: Changes in Circulating Serum Estradiol
Description: Circulating serum estradiol pre and post treatment to determine the effect of daily dose of 25mg of exemestane for 21-42 days.
Time Frame: Baseline up to 2 months
Population: Site did not collect data on the 3 participants omitted from the count
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment (Exemestane)
Number analyzed (Participants) | 37
pg/mL | 4.08 (13.81)

3. Secondary Outcome: Changes in Circulating Serum Progesterone
Description: Circulating serum progesterone pre and post treatment to determine the effect of daily dose of 25mg of exemestane for 21-42 days.
Time Frame: Baseline up to 2 months
Population: Site did not collect the relevant information for the omitted 3 participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment (Exemestane)
Number analyzed (Participants) | 37
ng/mL | 0.22 (0.27)

4. Secondary Outcome: Percent of Participants by Pathological Response Class at 2 Months
Description: This measure assesses change in categories in pathological response. As pathological response is an ordered categorical variable with classes of No visible lesion, CAH/EIN, Grade I, Grade II, and Grade III in this study, a change in class from baseline to time of surgery represents a decrease or increase in disease severity.
Time Frame: Up to 2 months
Measure: Number; unit: Percent of participants
Arm/Group | Treatment (Exemestane)
Number analyzed (Participants) | 40
Percent of participants
  No visible lesion | 2.5
  CAH/EIN | 20
  Grade I (Low) EC | 57.5
  Grade II (Low) EC | 10
  Grade III (High) EC | 10

5. Secondary Outcome: Change From Baseline in Percent of Cells Positive for Tissue Markers
Description: Assessment of change from baseline for apoptosis (cleaved caspase 3), proliferation (cyclin D1), insulin pathway (pAKT, IGF-1R), and endocrine regulation (estrogen receptor/progesterone receptor/androgen receptor). The units for absolute change in is % Positive.
Time Frame: Up to 2 months
Population: N=37 for caspase because there was not enough tissue on slide for 2 and 1 block was not sent. N=36 for cyclin D1 because 3 were missing data and 1 block was not sent. N=35 for pAKT because 3 were missing data, 1 did not have enough tissue, and 1 block was not sent. N=22 for IGF-1R because 1 black was not sent, 5 did not have enough tissue, and the rest are missing data.
Measure: Mean (Standard Deviation); unit: % positive
Arm/Group | Treatment (Exemestane)
Number analyzed (Participants) | 37
% positive
  Cleaved capsase | -0.17 (0.18)
  Cyclin D1: number analyzed (Participants) | 36
  Cyclin D1 | -0.07 (0.22)
  pAKT: number analyzed (Participants) | 35
  pAKT | -0.12 (0.27)
  IGF-1R: number analyzed (Participants) | 22
  IGF-1R | -2.50 (3.00)

6. Secondary Outcome: Deoxyribonucleic Acid (DNA) Mutational Analysis
Description: Will be analyzed by next generation sequencing.
Time Frame: Up to 2 months
Population: Samples were collected from participants. After enrollment was completed, the intended laboratory was no longer available to process the samples. There are no data to report and there is no intent to analyze these samples in the future.
Measure: Number; unit: percentage of cells
Arm/Group | Treatment (Exemestane)
Number analyzed (Participants) | 22
percentage of cells | NA — Samples were collected from participants. After enrollment was completed, the intended laboratory was no longer available to process the samples. There are no data to report.

7. Secondary Outcome: Protein Markers
Description: Perform pre- and post-treatment proteomic analysis of vaginal proteins from tampon recovery to identify biomarkers that may predict response to exemestane treatment.
Time Frame: Up to 2 months
Population: Tampon submission was optional and not all participants submitted tampon samples.
Measure: Number; unit: number of proteins
Arm/Group | Treatment (Exemestane)
Number analyzed (Participants) | 22
number of proteins | 85

8. Secondary Outcome: Ki-67 Expression With Historic Controls
Description: Will compare Ki-67 expression between participants samples and historically matched samples.
Time Frame: Up to 2 months
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Treatment (Exemestane)
Number analyzed (Participants) | 40
percentage of cells | -0.07 (0.10)

9. Secondary Outcome: Plasma Levels of Exemestane
Description: Will evaluate plasma levels of exemestane pre and post treatment.
Time Frame: Up to 2 months
Population: 40th specimen was not collected by the site.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment (Exemestane)
Number analyzed (Participants) | 39
ng/mL | 2.51 (1.23)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Treatment (Exemestane)
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 38/40
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Exemestane) (N=40)
Hot flashes (Vascular disorders) | 21
Hypertension (Vascular disorders) | 17
Flushing (Vascular disorders) | 1
Diarrhea (Gastrointestinal disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Bloating (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Blurred vision (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 8
Dizziness (Nervous system disorders) | 4
Concentration impairment (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Fatigue (General disorders) | 9
Edema limbs (General disorders) | 4
Chills (General disorders) | 1
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Alanine aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Urinary frequency (Renal and urinary disorders) | 2
Urinary urgency (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT03300557/Prot_SAP_000.pdf